CLINICAL TRIAL: NCT06078865
Title: FX Shoulder Post-Market Follow-Up Clinical Study
Brief Title: FX Shoulder Prospective Clinical Study
Status: Recruiting | Type: Observational
Sponsor: FX Shoulder Solutions (Industry)
Responsible Party: Sponsor
Other Study IDs: FXShoulder2020-01; FXShoulder2020-1 (Other: FX Shoulder Solutions)
Record Dates: First submitted 2023-09-26; First posted 2023-10-12 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Osteoarthritis Shoulder; Rotator Cuff Syndrome of Shoulder and Allied Disorders; Fracture, Shoulder
Keywords: Osteoarthritis; Fracture; rotator cuff tear; shoulder trauma
MeSH Terms: conditions — Shoulder Fractures; Osteoarthritis; Fractures, Bone; Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Subjects: Subjects implanted with the shoulder replacement medical devices manufactured by FX Shoulder Solutions
  Interventions: Device: FX Artificial Shoulder Prosthesis

INTERVENTIONS:
Device: FX Artificial Shoulder Prosthesis — Humelock II Anatomic Shoulder System, Humelock II Reversible Shoulder System, Humelock Reverse Shoulder System, Humeris Shoulder System, Easytech Anatomical Shoulder System, FXV135 Mini Shoulder System, FXV135 Humelock Shoulder System

SUMMARY:
Prospective Multi-Center Registry on study subjects with implanted devices marketed and legally commercialized in the USA by FX Shoulder Solutions.

DETAILED DESCRIPTION:
To evaluate patient outcomes following shoulder replacement with FX Shoulder Solutions medical devices and demonstrate effectiveness, safety and survivorship of FX Shoulder Solutions medical devices.

To provide data and analysis to FX Shoulder Solutions to meet regulatory requirements.

To provide data and analysis for presentations, abstracts, publications and other public release of results.

A patient is considered a success at minimum of 2 years post-operative follow-up based upon the following composite clinical success (CCS):

* Adjusted Constant Score that is ≥ 54 and improvement of ≥ 10 points from baseline
* No continuous radiolucency or device migration/subsidence
* No revision surgery
* No serious device related adverse event

The Registry will continue to follow patients to 10 years post-operative to track survivorship.

ELIGIBILITY:
Inclusion Criteria:

Receive an FX shoulder replacement medical device in accordance with the Indications for Use for the selected device system.

Exclusion Criteria:

Patient who does not meet the inclusion criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects implanted with the shoulder replacement medical devices manufactured by FX Shoulder Solutions and distributed by FX Shoulder Solutions
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2021-03-31 (Actual); Primary Completion 2031-12-30 (Estimated); Study Completion 2031-12-30 (Estimated)

PRIMARY OUTCOMES:
A patient is considered a success at post-operative follow-up based upon the following composite clinical success (CCS): | 2 years
  Adjusted Constant Score that is ≥ 54 and improvement of ≥ 10 points from baseline.
  No continuous radiolucency or device migration/subsidence No revision surgery No serious device related adverse event.
Survivorship | 10 years
  Follow patient's post-operative to track survivorship.

SECONDARY OUTCOMES:
Adjusted Constant Score | 6 weeks, 3, 6, 12, and 24 months.
  The Constant-Murley score (CMS) is a validated 100-points scale composed of a number of individual parameters. These parameters define the level of pain and the ability to carry out the normal daily activities of the patient. The test is divided into four subscales: pain (15 points), activities of daily living (20 points), strength (25 points) and range of motion (40 points) with the subject completing the assessment prior to the Investigator completing their part of the assessment. The higher the score, the higher the quality of the function.
  An Adjusted Constant score will be calculated using normalized values to account for age and gender, as based upon anatomical gender at birth.
QuickDASH | 6 weeks, 3, 6, 12, and 24 months.
  QuickDASH measures an individual's ability to complete tasks, absorb forces, and severity of symptoms.
  The QuickDASH tool uses a 5-point Likert scale from which the patient can select an appropriate number corresponding to his/her severity level/ function level. The higher the score, the higher the function and lower pain in the patient.
American Shoulder and Elbow Surgeon (ASES) | 6 weeks, 3, 6, 12, and 24 months
  ASES is a validated patient-reported outcome which is composed of 10 functional questions and one pain VAS. The total score is of 100 maximum points and weighted evenly between pain and function
Visual Analog Scale (VAS). | 6 weeks, 3, 6, 12, and 24 months
  A validated measurement of pain in a patient where 0 indicates no pain and 100 indicates severe pain. The VAS is a straight horizontal line of fixed length.
Range of Motion (ROM) | 6 weeks, 3, 6, 12, and 24 months
  The patient performs active movements in all functional planes for the shoulder. Includes flexion, extension, abduction, adduction and internal and external rotation. Investigator estimates the range of movement and compares the affected with the unaffected shoulder and the normal expected range.
Secondary Surgical Interventions (SSI) | 24 months and at 5 years postoperative
  SSI's are re-operations, revisions, and removals.
Serious Adverse Event | 24 months and at 5 years postoperative
  1. Led to a death.
  2. Resulted in life threatening illness or injury.
  3. Resulted in patient hospitalization or prolongation of existing hospitalization.
  4. Resulted in patient disability or permanent damage or required intervention to prevent permanent impairment/damage.
  5. Led to a congenital abnormality or birth defect.
Serious Adverse Device Effects (SADE) | 24 months and at 5 years postoperative.
  Adverse device effect that has resulted in any of the consequences characteristic of a serious adverse event.
Radiographic Reviews and Assessments. | 24 months and at 5 years postoperative.
  Monitor implant integrity and signs of implant loosening.
Survival | 24 months and at 5 years
  Subject disposition.

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Trier, PhD, Study Director — FX Shoulder Solutions
Locations (4):
- United States (4):
  - OrthoArizona, Gilbert, Arizona
  - First Settlement Orthopedics, Marietta, Ohio
  - Orthopedics Rhode Island, Wakefield, Rhode Island
  - Texas Orthopedic Specialists, Bedford, Texas

IPD SHARING:
Plan to Share IPD: No